CLINICAL TRIAL: NCT01240538
Title: A Phase 1 Dose Escalation Study of Reolysin, a Replication Competent Reovirus, in Pediatric Patients With Relapsed or Refractory Solid Tumors
Brief Title: Viral Therapy in Treating Young Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02617; NCI-2011-02617 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688938; ADVL1014 (Other: COG Phase I Consortium); ADVL1014 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: interventions — reolysin; Cyclophosphamide

ARMS (1):
- Treatment (virus and chemotherapy) (Experimental): Patients receive wild-type reovirus IV over 60 minutes QD on days 1-5. Some patients also receive cyclophosphamide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: wild-type reovirus; Drug: cyclophosphamide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: wild-type reovirus — Given IV
  Other Names: REOLYSIN
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and the best dose of viral therapy in treating young patients with solid tumors that have come back or that have not responded to standard therapy. Some tumors have cells with a genetic weakness that makes them unable to fight off a virus called wild-type reovirus. The virus causes cells with this weakness to die, and may therefore be able to kill tumor cells without damaging normal cells. Cyclophosphamide is a drug used in chemotherapy that stops tumor cells from dividing and causes them to die. Giving wild-type reovirus together with cyclophosphamide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of REOLYSIN (wild-type reovirus) administered as an intravenous infusion daily for 5 days, every 28 days to children with relapsed or refractory solid tumors.

II. To define and describe the toxicities of Reolysin in these patients. III. To define the toxicity and tolerability of combining Reolysin with oral cyclophosphamide in these patients.

IV. To characterize the pharmacokinetics (time course of viral clearance) of Reolysin in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To define the antitumor activity of Reolysin within the confines of a phase I study.

II. To evaluate the development of neutralizing antibodies to Reolysin following intravenous administration of Reolysin alone and in combination with cyclophosphamide.

III. To assess the biologic activity of Reolysin.

OUTLINE: This is a dose-escalation study of wild-type reovirus.

Patients receive wild-type reovirus intravenously (IV) over 60 minutes once daily (QD) on days 1-5. Some patients also receive cyclophosphamide orally (PO) on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory solid tumors, with the exception of central nervous system (CNS) tumors and lymphomas, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50 for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy and immunizations
* Must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
* At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines
* At least 3 half-lives of the antibody after the last dose of a monoclonal antibody
* >= 2 weeks for local palliative radiation therapy (XRT) (small port); >= 24 weeks must have elapsed if prior total-body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* No evidence of active graft vs host disease and >= 12 weeks must have elapsed since stem cell transplant or infusion
* Patients must not have received any previous viral-based anti-neoplastic therapies
* Viral immunizations, including influenza, may not have been administered within 7 days prior to enrollment; Note: patients may not receive any viral immunizations after enrolling on study until 28 days post their last planned REOLYSIN infusion
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3 (transfusion independent (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study but not evaluable for hematologic toxicity (maximum of one per cohort); such patients must meet the blood counts above (may receive transfusions provided they are not be known to be refractory to red cell or platelet transfusion); if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min OR serum creatinine based on age and/or gender as follows:

  * 0.8 mg/dL (3 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Bilirubin (sum of conjugated plus unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Shortening fraction >= 27% by echocardiogram OR ejection fraction >= 50% by gated radionuclide study
* Normal pulmonary function tests (PFTs) (including diffusion capacity of carbon monoxide [DLCO]) if there is clinical indication for determination (e.g. dyspnea at rest, known requirement for supplemental oxygen); for patients who do not have respiratory symptoms, full PFTs are NOT required
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4 (CTCAE v. 4) resulting from prior therapy must be =< grade 2
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients who have an uncontrolled infection are not eligible
* Patients with chronic diarrhea, urinary incontinence during the day or at night, or patients who are not completely toilet trained will not be eligible
* Patients will be excluded if they have household contacts who are pregnant, immunosuppressed or infants less than 3 months of age; household contacts are defined as anyone living with the patient during the isolation period of the treatment cycles
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with known human immunodeficiency virus (HIV) or hepatitis B or C are excluded due to risk of viral infectivity of REOLYSIN; therefore, patients with a pre-existent infection are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post transplant are not eligible for this trial
* Patients must not have received corticosteroids, immune modulators or antiviral therapy for 7 days prior to enrollment and must not have an anticipated need for any of these therapies, intravenous immune globulin (IVIG) must not have been administered within 2 weeks prior to enrollment
* Patients should avoid taking acetaminophen with REOLYSIN; whenever suitable, physicians should utilize alternative medications
* Patients with known germline mutations affecting Ras activation (e.g. NF-1, Cardio-facial-cutaneous syndrome, Noonan syndrome, Costello syndrome) will be excluded from enrollment
* Patients with known metastatic CNS disease involvement are excluded
* Patients with primary CNS tumors are excluded

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD), defined as the maximum dose at which fewer than one-third of patients experience dose-limiting toxicity (DLT), graded using the NCI CTCAE v. 4.0 | Up to 28 days

SECONDARY OUTCOMES:
Time course of viral clearance of wild-type reovirus | Up to 3 months
  Summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Development of neutralizing antibodies to wild-type reovirus | Up to 3 months
  Summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Disease response, assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 1 year
  Will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: E. Anders Kolb, Principal Investigator — COG Phase I Consortium
Locations (27):
- United States (25):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Childrens Hospital of Orange County, Orange, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec